CLINICAL TRIAL: NCT00994838
Title: Reduced Calorie Diet Intervention in Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kelly Birdwell, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091030
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- reduced calorie diet (Active Comparator): 10% reduction in total daily calories (≈ 300 kcal reduction) from carbohydrates and fat from the usual daily energy consumption
  Interventions: Other: reduced calorie diet
- standard diet (No Intervention)

INTERVENTIONS:
Other: reduced calorie diet — 10% reduction in total daily calories (≈ 300 kcal reduction) from carbohydrates and fat from the usual daily energy consumption
  Arms: reduced calorie diet

SUMMARY:
The purpose of this study is to measure the effect of a reduced calorie diet intervention in new kidney transplant recipients on the outcomes weight gain, oxidative stress, and insulin resistance.

DETAILED DESCRIPTION:
Kidney transplantation is the preferred renal replacement therapy for end stage renal disease (ESRD) because it affords survival and quality of life advantages over maintenance dialysis.1 The number of transplants performed increases each year, with currently over 150,000 individuals living in the United States with a kidney transplant. This is in the setting of 68,000 patients on the wait list with a median wait time of 4 years for an available organ.2 Despite the survival benefit over dialysis, transplanted patients still have a greatly increased risk of cardiovascular disease (CVD) over the general population, and CVD is the leading cause of death among recipients with a functioning graft.3 Given the long wait times for kidneys due to organ shortage, extensive resources used, and support needed for each transplant procedure, it is imperative that we improve long term patient and graft survival. Accordingly, modification of CVD risk profile is of paramount importance in kidney transplant patients.

The etiology of increased risk of CVD in kidney transplant patients is multi-factorial and includes the high burden of CVD and its risk factors present prior to transplant, as well as increasing prevalence of these risk factors in the post transplant period due to transplant associated weight gain, immunosuppression side effects, metabolic consequences of a functioning kidney, and allograft dysfunction. Efforts to reduce CVD risk factors have yet to be adequately implemented and rigorously studied in the kidney transplant population.

Obesity at the time of transplant is common and associated with several CVD risk factors post transplant, including hypertension, hyperlipidemia, diabetes mellitus, metabolic syndrome, and inflammation. Obesity is also associated with potentially poorer graft outcomes, including death censored graft loss and chronic allograft failure.4 In addition, the majority of patients gain weight post transplantation, primarily in the form of fat mass. Post transplant weight gain is also associated with increased prevalence of known CVD risk factors, CVD death, and graft loss.5 The increased burden of CVD in kidney transplant patients makes obesity prevention and treatment strategies appealing interventions to improve long-term outcomes, both in terms of graft and overall survival. In this study we will measure the effect of a low calorie diet intervention in new kidney transplant recipients on the outcomes weight gain, oxidative stress, and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 65 years;
* BMI 25 to 40 kg/m2;
* First time kidney transplant;
* Single organ transplant;
* Ability to understand and voluntarily provide informed consent.

Exclusion Criteria:

* Type 1 DM;
* Type 2 DM on diabetic medications/insulin;
* Biopsy proven acute rejection in the first 3 months post transplant;
* Active coronary disease;
* Immunosuppressive therapy at time of transplant (use prior to what is given for transplant procedure);
* Atrial fibrillation (only for those undergoing the optional Pulse Wave Velocity);
* Hypersensitivity to organic nitrates, isosorbide, or nitroglycerin (only for those undergoing the optional brachial artery Doppler).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
a significant improvement in measures of body composition (including weight, BMI, and fat mass) | 12 months

SECONDARY OUTCOMES:
an improvement in insulin resistance | 12 months
a decrease in oxidative stress markers | 12 months
an improvement in kidney function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelly A Birdwell, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States